CLINICAL TRIAL: NCT07376837
Title: Evaluating the Feasibility, Safety and Efficacy of Radiofrequency Ablation (RFA) for Curative Treatment of Small Low-Risk Thyroid Papillary Cancer: A Pilot Single Arm Clinical Trial
Brief Title: Radiofrequency Ablation for Curative Treatment of Small Low-Risk Papillary Thyroid Cancer: Pilot Study
Acronym: PTC-RFA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-5017
Record Dates: First submitted 2026-01-15; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Papillary Carcinoma
Keywords: Thyroid Radiofrequency Ablation; Minimally Invasive Treatment; Thyroid Papillary Carcinoma; Ultrasound-guided; Low-risk cancer-focused; Thyroid-sparing
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, single-arm interventional pilot study designed to evaluate radiofrequency ablation (RFA) as a curative-intent treatment for small, low-risk papillary thyroid cancer. All enrolled participants receive the same intervention (RFA), with no randomization or comparison group, as the primary purpose is to assess feasibility, safety, and preliminary effectiveness rather than comparative efficacy.
  Participants undergo a one-time ultrasound-guided RFA procedure, followed by a structured follow-up schedule over 12 months that includes clinical assessments, imaging, laboratory testing, voice evaluations, patient-reported outcome measures, and a biopsy of the treated site at 6-12 months to assess local cancer control. Outcomes are collected prospectively using standardized protocols.
  As a pilot study, this model is intended to generate high-quality preliminary data to inform the design of future larger, potentially randomized studies comparing RFA with stand
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiofrequency Ablation (RFA) for Low-Risk Papillary Thyroid Cancer (Experimental): This single study arm includes adult participants with biopsy-confirmed, low-risk papillary thyroid cancer (<2 cm) who undergo curative-intent radiofrequency ablation (RFA) of the thyroid tumor. RFA is performed once, on an outpatient basis, using a percutaneous, ultrasound-guided approach with an internally cooled radiofrequency electrode. The procedure is carried out under local anesthesia with conscious sedation, using a standardized moving-shot technique, with hydrodissection as needed to protect adjacent structures.
  No study drugs are administered as part of this intervention. The RFA procedure is a one-time treatment, although repeat ablation may be considered if residual disease is identified during follow-up, based on clinical judgment and participant consent.
  All participants in this arm follow the same post-procedure monitoring and follow-up schedule, which includes clinical assessments, neck ultrasound, thyroid blood tests, voice evaluation, patient-reported outcome quest
  Interventions: Procedure: Radiofrequency Ablation of Papillary Thyroid Cancer; Device: VIVA combo RF Generator with Coagulation Electrode

INTERVENTIONS:
Procedure: Radiofrequency Ablation of Papillary Thyroid Cancer — Radiofrequency ablation (RFA) is a minimally invasive, image-guided procedure used to destroy targeted thyroid cancer tissue using controlled heat. In this study, RFA is performed percutaneously under real-time ultrasound guidance using an internally cooled radiofrequency electrode inserted into the thyroid tumor through the skin. The procedure is carried out under local anesthesia with conscious sedation.
  A standardized moving-shot technique is used to ablate the entire tumor, and hydrodissection may be applied to protect nearby critical structures such as the vocal cord nerve, trachea, and esophagus. RFA is delivered as a single-session treatment with curative intent and is performed on an outpatient basis, with most patients returning home the same day.
  This intervention preserves the thyroid gland and avoids surgical incisions. Treatment response is assessed through follow-up imaging, clinical evaluations, patient-reported outcomes, and an ultrasound-guided biopsy of the treated
Device: VIVA combo RF Generator with Coagulation Electrode — Evaluating the Feasibility, Safety and Efficacy of Radiofrequency Ablation (RFA) for Curative Treatment of Small Low-Risk Thyroid Papillary Cancer: A Pilot Single Arm Clinical Trial - VIVA combo RF Generator with Coagulation Electrode
  Other Names: Southmedic Inc,

SUMMARY:
This pilot, single-arm clinical study evaluates the feasibility, safety, and effectiveness of radiofrequency ablation (RFA) as a curative treatment for small, low-risk papillary thyroid cancer (PTC). The study will enroll 30 adult patients (≥18 years) with biopsy-confirmed PTC measuring <2 cm, who decline surgery or active surveillance, or who are transitioning from active surveillance to active treatment.

Eligible participants will undergo ultrasound-guided RFA performed with curative intent at University Health Network. Patients will be followed for up to 12 months with scheduled clinical visits, neck ultrasounds, blood tests, voice assessments, and patient-reported outcome questionnaires. A biopsy of the ablation site at 6-12 months will be used to assess local cancer control.

The primary objective is to determine the local cure rate and safety profile of RFA for low-risk PTC. Secondary objectives include evaluating post-ablation ultrasound features, patient-reported quality of life, and the feasibility of implementing a multidisciplinary thyroid RFA program within routine clinical practice.

Results from this study will provide important preliminary data to inform future larger trials comparing RFA with surgery and active surveillance for selected patients with low-risk papillary thyroid cancer.

DETAILED DESCRIPTION:
This study is a pilot clinical trial designed to evaluate a less invasive treatment option for adults with small, low-risk papillary thyroid cancer (PTC). PTC is the most common type of thyroid cancer and is often slow growing with an excellent prognosis. Standard treatment usually involves surgery to remove part or all of the thyroid gland. While surgery is highly effective, it may be associated with complications such as voice changes, low calcium levels, prolonged recovery, and the need for lifelong thyroid hormone replacement. For some patients, close monitoring without treatment (active surveillance) is an option, but this approach can cause ongoing anxiety and uncertainty.

Radiofrequency ablation (RFA) is a minimally invasive, image-guided procedure that uses controlled heat to destroy targeted tissue. RFA has been widely used to treat benign thyroid nodules and is increasingly being explored as a treatment for carefully selected small thyroid cancers. This study aims to determine whether RFA can safely and effectively eliminate small PTCs while preserving the thyroid gland and reducing the impact of treatment on patients' daily lives.

The study will enroll 30 adult participants (18 years or older) with biopsy-confirmed papillary thyroid cancer measuring less than 2 cm, with no evidence of spread outside the thyroid or to lymph nodes. All participants will have previously been offered standard treatment options and have chosen not to undergo surgery or active surveillance, or will be transitioning from active surveillance to active treatment. Each potential participant will be reviewed by a multidisciplinary team that includes radiology, endocrinology, and surgical specialists to ensure the treatment is appropriate and safe.

The RFA procedure will be performed on an outpatient basis under local anesthesia and light sedation, using real-time ultrasound guidance to precisely target the cancer while protecting nearby structures such as the vocal cords, trachea, and esophagus. Patients are typically observed briefly after the procedure and can return home the same day.

Following treatment, participants will be followed closely for up to 12 months. Follow-up includes clinic visits, neck ultrasound examinations, blood tests to assess thyroid function, voice assessments, and questionnaires that evaluate symptoms, quality of life, satisfaction with treatment, and decision-related concerns. A key component of follow-up is an ultrasound-guided biopsy of the treated area performed 6 to 12 months after RFA, which will be used to determine whether the cancer has been successfully eradicated.

The primary focus of the study is to assess local cancer control and safety of RFA, including the frequency and severity of any complications. Additional goals include understanding how treated thyroid cancers appear on ultrasound over time, evaluating patient-reported outcomes, and assessing the practicality of delivering and sustaining a multidisciplinary thyroid RFA program within a Canadian academic health-care setting.

The results of this study will provide important early evidence on the role of radiofrequency ablation as a potential alternative to surgery for selected patients with low-risk papillary thyroid cancer and will help guide future larger clinical trials and treatment guidelines.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed papillary thyroid carcinoma (PTC) by fine-needle aspiration (FNA -Bethesda V/VI ) or core needle biopsy.
* Single or multiple lesions, each 2.0 cm in maximum diameter.
* Intrathyroidal tumors (i.e., no extrathyroidal extension, no clinical/radiological evidence of nodal metastases, nor distant metastases).
* Lesions located at a safe distance (>2 mm) from critical structures (e.g., trachea, esophagus, carotid artery) or accessible with hydrodissection.
* ≤T1b (i.e. < 2cm maximal diameter), N0 or Nx, M0 (no clinical or radiological evidence of lymph node or distant metastasis).
* Patients unfit for surgery due to comorbidities or who refuse surgery.
* ≥18 years old
* Not pregnant at the time of RFA.
* Able to understand and voluntarily sign informed consent.

Exclusion Criteria:

* Evidence of lymph node involvement (clinically or radiologically suspicious or confirmed metastatic nodes) or distant metastasis (e.g., lung, bone).
* Tumors with extrathyroidal extension
* Tumors with extensive calcification
* Tumors located within 2 mm of critical structures where RFA would pose an unacceptably high risk and where hydrodissection is not feasible.
* Previous thyroid surgery or ablation (RFA, ethanol, laser, or microwave) at the index tumor site.
* Known diagnosis of anaplastic, poorly differentiated, or other aggressive thyroid cancer variants.
* Pregnant or breastfeeding at the time of enrollment.
* Bleeding diathesis or use of anticoagulants that cannot be discontinued safely prior to RFA.
* Severe comorbid illness that limits life expectancy to less than 5 years.
* Inability to adhere to study follow-up schedule or procedures or lacking decision-making capacity.
* Implanted electrical devices such as pacemakers or neurostimulators
* Infection in the neck including skin infection or thyroiditis at time of planned ablation.
* Severe cervical anatomy distortion (prior neck surgery or radiation with distorted anatomy that prevents safe RFA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Local Cure Rate of Papillary Thyroid Cancer (PTC) following Radiofrequency | From enrollment to the end of treatment at 12 months.
  Local cure rate of papillary thyroid cancer (PTC) following radiofrequency ablation, assessed by ultrasound-guided fine needle aspiration or core biopsy of the ablation site at 6-12 months, with local cure defined as no evidence of malignancy on biopsy (when diagnostic material is obtained).
Safety of the RFA procedure | From enrollment to the end of treatment at 12 months.
  Safety of the RFA procedure, measured by the incidence and nature of procedure-related complications, including but not limited to voice changes, hematoma, pain, skin burns, and other adverse events.

SECONDARY OUTCOMES:
Ultrasound characteristics following RFA | From enrollment to the end of treatment at 12 months
  including features used to differentiate successfully treated tumors from residual or recurrent disease
Tumor volume change over time, | at 6 and 12 months post-RFA
  measured by volume reduction ratio (VRR)
Complication rate of radiofrequency ablation, including but not limited to: | From Treatment to the end of study at 12 months
  Voice changes, Hematoma, Pain, and Skin burns
Patient-reported outcome (Patient Satisfaction) | From enrollment to the end of study at 12 months.
  Patient satisfaction will be assessed using a study-specific questionnaire evaluating satisfaction with the procedure and overall care. Scores range from 1 to 5, with higher scores indicating greater satisfaction (better outcome) and lower scores indicating lower satisfaction.
Patient-reported outcome Voice Handicap Index-10 (VHI-10) | Time Frame: From enrollment to the end of study at 12 months.
  Self-reported Voice Handicap Index-10 (VHI-10): Total score range 0-40; higher scores indicate worse voice-related handicap.
Patient-reported outcome (EORTC QLQ-C30) | From enrollment to the end of the study at 12 months
  The EORTC QLQ-C30 is a validated cancer-specific questionnaire assessing global health status and multiple functional and symptom domains. Scores are transformed to a 0-100 scale. For functional and global health status scales, higher scores indicate better quality of life/functioning, whereas for symptom scales, higher scores indicate worse symptom burden.
Patient Reported outcome - The Assessment of Survivor Concerns (ASC) | From enrollment to the end of study at 12 months
  The Assessment of Survivor Concerns (ASC) is a validated patient-reported questionnaire designed to evaluate cancer survivors' concerns across multiple domains (e.g., physical, emotional, social, and existential concerns). Total scores range from 0 to 100, with higher scores indicating greater survivor concerns (worse outcomes) and lower scores indicating fewer concerns (better outcomes).
Patient-Reported Outcome - Decision Regret Scale (DRS) | From enrollment to the end of study at 12 months
  Decision regret will be assessed using the Decision Regret Scale (DRS), a validated patient-reported questionnaire measuring distress or remorse after a healthcare decision. Scores are transformed to a 0-100 scale, with higher scores indicating greater decision regret (worse outcome) and lower scores indicating less regret (better outcome).
Changes in thyroid biochemical markers over time, including: | From enrollment to the end of study at 12 months.
  Thyroid-stimulating hormone (TSH)
  Free T4 (if TSH abnormal)
  Thyroglobulin
  Thyroglobulin antibody levels

CONTACTS AND LOCATIONS:
Overall Officials: Sangeet Ghai, MD, Principal Investigator — University Health Network - Toronto General Hospital

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) from this study may be shared with qualified researchers upon reasonable request. Data sharing will be considered after completion of the primary analyses and publication of the main study results. Shared data will exclude all direct identifiers and will comply with institutional policies, REB requirements, and applicable privacy legislation.
  Requests will be reviewed by the study Principal Investigator to ensure scientific validity, ethical appropriateness, and alignment with the original consent. Data will be shared under a data-sharing agreement outlining the permitted use of the data, data security requirements, and restrictions on re-identification or further sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: De-identified IPD and supporting documents will be made available after publication of the primary study results or within 12 months of study completion, whichever occurs first.
Access Criteria: IPD will be shared upon reasonable request with qualified researchers. Requests must include a brief research proposal and intended use of the data. All requests will be reviewed and approved by the Principal Investigator and must comply with Research Ethics Board (REB) approval, participant consent, and institutional data-sharing policies.
  Conditions of use:
  Data will be provided in a de-identified format and shared under a formal data-sharing

REFERENCES:
- [Result] Sakai T, Sugitani I, Ebina A, Fukuoka O, Toda K, Mitani H, Yamada K. Active Surveillance for T1bN0M0 Papillary Thyroid Carcinoma. Thyroid. 2019 Jan;29(1):59-63. doi: 10.1089/thy.2018.0462. Epub 2019 Jan 8. PMID 30560718
- [Result] Dionisio T, Mauri G. Ultrasound Evaluation of Ablated Thyroid Nodules: An Emerging Problem. Thyroid. 2024 Aug;34(8):1062-1063. doi: 10.1089/thy.2024.0244. Epub 2024 Jul 4. No abstract available. PMID 38916184
- [Result] Gotay CC, Pagano IS. Assessment of Survivor Concerns (ASC): a newly proposed brief questionnaire. Health Qual Life Outcomes. 2007 Mar 13;5:15. doi: 10.1186/1477-7525-5-15. PMID 17352831
- [Result] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Result] Hawthorne G, Sansoni J, Hayes L, Marosszeky N, Sansoni E. Measuring patient satisfaction with health care treatment using the Short Assessment of Patient Satisfaction measure delivered superior and robust satisfaction estimates. J Clin Epidemiol. 2014 May;67(5):527-37. doi: 10.1016/j.jclinepi.2013.12.010. PMID 24698296
- [Result] Rosen CA, Lee AS, Osborne J, Zullo T, Murry T. Development and validation of the voice handicap index-10. Laryngoscope. 2004 Sep;114(9):1549-56. doi: 10.1097/00005537-200409000-00009. PMID 15475780
- [Result] Bresner L, Banach R, Rodin G, Thabane L, Ezzat S, Sawka AM. Cancer-related worry in Canadian thyroid cancer survivors. J Clin Endocrinol Metab. 2015 Mar;100(3):977-85. doi: 10.1210/jc.2014-3169. Epub 2014 Nov 13. PMID 25393643
- [Result] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Result] Singer S, Jordan S, Locati LD, Pinto M, Tomaszewska IM, Araujo C, Hammerlid E, Vidhubala E, Husson O, Kiyota N, Brannan C, Salem D, Gamper EM, Arraras JI, Ioannidis G, Andry G, Inhestern J, Gregoire V, Licitra L; EORTC Quality of Life Group, the EORTC Head and Neck Cancer Group, and the EORTC Endocrine Task Force. The EORTC module for quality of life in patients with thyroid cancer: phase III. Endocr Relat Cancer. 2017 Apr;24(4):197-207. doi: 10.1530/ERC-16-0530. Epub 2017 Feb 21. PMID 28223365
- [Result] Kim C, Lee JH, Choi YJ, Kim WB, Sung TY, Baek JH. Complications encountered in ultrasonography-guided radiofrequency ablation of benign thyroid nodules and recurrent thyroid cancers. Eur Radiol. 2017 Aug;27(8):3128-3137. doi: 10.1007/s00330-016-4690-y. Epub 2016 Dec 14. PMID 27975148
- [Result] Baek JH, Lee JH, Sung JY, Bae JI, Kim KT, Sim J, Baek SM, Kim YS, Shin JH, Park JS, Kim DW, Kim JH, Kim EK, Jung SL, Na DG; Korean Society of Thyroid Radiology. Complications encountered in the treatment of benign thyroid nodules with US-guided radiofrequency ablation: a multicenter study. Radiology. 2012 Jan;262(1):335-42. doi: 10.1148/radiol.11110416. Epub 2011 Oct 13. PMID 21998044
- [Result] Li X, Li Y, Yan L, Xiao J, Yang Z, Jing H, Zhang M, Luo Y. Sonographic Evolution and Pathologic Findings of Papillary Thyroid Cancer After Radiofrequency Ablation: A Five-Year Retrospective Cohort Study. Thyroid. 2024 Jan;34(1):54-63. doi: 10.1089/thy.2023.0415. Epub 2023 Nov 20. PMID 37885207
- [Result] Rachmasari KN, Schmitz JJ, Castro MR, Kurup AN, Lee RA, Stan MN. Exploring Radiofrequency Ablation for T1 Papillary Thyroid Cancer in the United States: Mayo Clinic Experience. Mayo Clin Proc. 2024 Nov;99(11):1702-1709. doi: 10.1016/j.mayocp.2024.04.010. Epub 2024 Aug 2. PMID 39093272
- [Result] Li X, Yan L, Xiao J, Li Y, Yang Z, Zhang M, Luo Y. Long-Term Outcomes and Risk Factors of Radiofrequency Ablation for T1N0M0 Papillary Thyroid Carcinoma. JAMA Surg. 2024 Jan 1;159(1):51-58. doi: 10.1001/jamasurg.2023.5202. PMID 37878294
- [Result] Zhang M, Luo Y, Zhang Y, Tang J. Efficacy and Safety of Ultrasound-Guided Radiofrequency Ablation for Treating Low-Risk Papillary Thyroid Microcarcinoma: A Prospective Study. Thyroid. 2016 Nov;26(11):1581-1587. doi: 10.1089/thy.2015.0471. Epub 2016 Aug 18. PMID 27445090
- [Result] Cho SJ, Baek SM, Na DG, Lee KD, Shong YK, Baek JH. Five-year follow-up results of thermal ablation for low-risk papillary thyroid microcarcinomas: systematic review and meta-analysis. Eur Radiol. 2021 Sep;31(9):6446-6456. doi: 10.1007/s00330-021-07808-x. Epub 2021 Mar 13. PMID 33713168
- [Result] Cho SJ, Suh CH, Baek JH, Chung SR, Choi YJ, Chung KW, Shong YK, Lee JH. Active Surveillance for Small Papillary Thyroid Cancer: A Systematic Review and Meta-Analysis. Thyroid. 2019 Oct;29(10):1399-1408. doi: 10.1089/thy.2019.0159. Epub 2019 Sep 27. PMID 31368412
- [Result] Sawka AM, Ghai S, Yoannidis T, Rotstein L, Gullane PJ, Gilbert RW, Pasternak JD, Brown DH, Eskander A, Almeida JR, Irish JC, Higgins K, Enepekides DJ, Monteiro E, Banerjee A, Shah M, Gooden E, Zahedi A, Korman M, Ezzat S, Jones JM, Rac VE, Tomlinson G, Stanimirovic A, Gafni A, Baxter NN, Goldstein DP. A Prospective Mixed-Methods Study of Decision-Making on Surgery or Active Surveillance for Low-Risk Papillary Thyroid Cancer. Thyroid. 2020 Jul;30(7):999-1007. doi: 10.1089/thy.2019.0592. Epub 2020 Apr 8. PMID 32126932
- [Result] Goldstein DP, Ghai S, Corsten M, Bissada E, Audet N, Zhang H, Nichols A, Morrison D, Johnson-Obeski S, Anderson DW, Prisman E, Baxter NN, Jones J, Gafni A, Witterick I, Sawka AM. Proceedings of the Canadian Thyroid Cancer Active Surveillance Study Group 2019 national investigator meeting. J Otolaryngol Head Neck Surg. 2021 Jun 25;50(1):40. doi: 10.1186/s40463-021-00514-0. PMID 34172096
- [Result] Sawka AM, Ghai S, Ihekire O, Jones JM, Gafni A, Baxter NN, Goldstein DP, On Behalf Of The Canadian Thyroid Cancer Active Surveillance Study Group. Decision-making in Surgery or Active Surveillance for Low Risk Papillary Thyroid Cancer During the COVID-19 Pandemic. Cancers (Basel). 2021 Jan 20;13(3):371. doi: 10.3390/cancers13030371. PMID 33498497
- [Result] Sawka AM, Ghai S, Rotstein L, Irish JC, Pasternak JD, Gullane PJ, Monteiro E, Gooden E, Brown DH, Eskander A, Zahedi A, Chung J, Su J, Xu W, Ihekire O, Jones JM, Gafni A, Baxter NN, Goldstein DP; Canadian Active Surveillance Study Group (Greater Toronto Area). A Quantitative Analysis Examining Patients' Choice of Active Surveillance or Surgery for Managing Low-Risk Papillary Thyroid Cancer. Thyroid. 2022 Mar;32(3):255-262. doi: 10.1089/thy.2021.0485. Epub 2022 Feb 17. PMID 35019770
- [Result] Sawka AM, Ghai S, Rotstein L, Irish JC, Pasternak JD, Monteiro E, Chung J, Zahedi A, Su J, Xu W, Jones JM, Gafni A, Baxter NN, Goldstein DP. Decision Regret Following the Choice of Surgery or Active Surveillance for Small, Low-Risk Papillary Thyroid Cancer: A Prospective Cohort Study. Thyroid. 2024 May;34(5):626-634. doi: 10.1089/thy.2023.0634. Epub 2024 Apr 8. PMID 38481111
- [Result] Ghai S, Goldstein DP, Sawka AM. Ultrasound Imaging in Active Surveillance of Small, Low-Risk Papillary Thyroid Cancer. Korean J Radiol. 2024 Aug;25(8):749-755. doi: 10.3348/kjr.2024.0148. Epub 2024 Jul 15. PMID 39028013
- [Result] Sawka AM, Ghai S, Rotstein L, Irish JC, Pasternak JD, Gullane PJ, Monteiro E, Zahedi A, Gooden E, Eskander A, Chung J, Devon K, Su J, Xu W, Jones JM, Gafni A, Baxter NN, Goldstein DP; Canadian Thyroid Cancer Active Surveillance Study Group (Greater Toronto Area). Gender Differences in Fears Related to Low-Risk Papillary Thyroid Cancer and Its Treatment. JAMA Otolaryngol Head Neck Surg. 2023 Sep 1;149(9):803-810. doi: 10.1001/jamaoto.2023.1642. PMID 37410454
- [Result] Ghai S, O'Brien C, Goldstein DP, Sawka AM; Canadian Thyroid Cancer Active Surveillance Study Group. Ultrasound in active surveillance for low-risk papillary thyroid cancer: imaging considerations in case selection and disease surveillance. Insights Imaging. 2021 Sep 16;12(1):130. doi: 10.1186/s13244-021-01072-9. PMID 34529219
- [Result] Sawka AM, Ghai S, Tomlinson G, Baxter NN, Corsten M, Imran SA, Bissada E, Lebouef R, Audet N, Brassard M, Zhang H, Gupta M, Nichols AC, Morrison D, Johnson-Obeski S, Prisman E, Anderson D, Chandarana SP, Ghaznavi S, Jones J, Gafni A, Matelski JJ, Xu W, Goldstein DP; Canadian Thyroid Cancer Active Surveillance Study Group. A Protocol for a Pan-Canadian Prospective Observational Study on Active Surveillance or Surgery for Very Low Risk Papillary Thyroid Cancer. Front Endocrinol (Lausanne). 2021 Jun 10;12:686996. doi: 10.3389/fendo.2021.686996. eCollection 2021. PMID 34194396
- [Result] Sawka AM, Ghai S, Tomlinson G, Rotstein L, Gilbert R, Gullane P, Pasternak J, Brown D, de Almeida J, Irish J, Chepeha D, Higgins K, Monteiro E, Jones JM, Gafni A, Goldstein DP. A protocol for a Canadian prospective observational study of decision-making on active surveillance or surgery for low-risk papillary thyroid cancer. BMJ Open. 2018 Apr 12;8(4):e020298. doi: 10.1136/bmjopen-2017-020298. PMID 29654030

DOCUMENTS (1):
  • Informed Consent Form (2026-01-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT07376837/ICF_000.pdf